CLINICAL TRIAL: NCT00297492
Title: Gradual vs. Abrupt Cessation Treatment for Smoking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, John Hughes, Professor of Psychiatry, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA011557-07 (NIH); R01DA011557-07 (NIH)
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Tobacco
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gradual reduction (Experimental): Intervention: Reduction Phone Counseling. Intervention: Pre-Quit Nicotine Lozenges. Intervention: Post-Quit Nicotine Lozenges.
  Interventions: Behavioral: Reduction Phone Counseling; Drug: Pre-Quit Nicotine Lozenges; Drug: Post-Quit Nicotine Lozenges
- Abrupt cessation (Active Comparator): Intervention: Abrupt Phone Counseling. Intervention: Post-Quit Nicotine Lozenges.
  Interventions: Behavioral: Abrupt Phone Counseling; Drug: Post-Quit Nicotine Lozenges
- Minimal intervention (Active Comparator): Intervention: Minimal Abrupt Phone Counseling. Intervention: Post-Quit Nicotine Lozenges.
  Interventions: Behavioral: Minimal Abrupt Phone Counseling; Drug: Post-Quit Nicotine Lozenges

INTERVENTIONS:
Behavioral: Reduction Phone Counseling — Counseling of smokers to undergo gradual reduction in cigarettes per day prior to quit date. This includes 5 counseling calls: 3 calls focused on reduction prior to the quit date, 1 call two days prior to the quit date to discuss common strategies for preparing to quit, and 1 call two days after the quit date to discuss relapse prevention. Telephone counseling also discusses the proper use of nicotine lozenges during reduction and after the quit date.
  Arms: Gradual reduction
Behavioral: Abrupt Phone Counseling — Counseling of smokers to set a quit date and not change cigarettes per day prior to quit date. This includes 5 counseling calls: 1 to set a quit date, 1 two days prior to the quit date to discuss common strategies for preparing to quit, and 3 after the quit date to discuss relapse prevention. Telephone counseling also discusses the proper use of nicotine lozenges after the quit date.
  Arms: Abrupt cessation
Behavioral: Minimal Abrupt Phone Counseling — Minimal counseling to mimic intervention at a primary care office. This includes 2 counseling calls: 1 to set a quit date and 1 two days after the quit date to discuss relapse prevention. Telephone counseling also discusses the proper use of nicotine lozenges after the quit date.
  Arms: Minimal intervention
Drug: Pre-Quit Nicotine Lozenges — 2 mg lozenges for participants usually smoke their first cigarette more than 30 minutes after awaking.
  4 mg lozenge for participants who usually smoke their first cigarette less than 30 minutes after awaking.
  Replace each forgone cigarette during reduction with one lozenge. Use additional lozenges to combat cravings to smoke.
  Other Names: Commit Nicotine Lozenges
  Arms: Gradual reduction
Drug: Post-Quit Nicotine Lozenges — 2 mg lozenges for participants usually smoke their first cigarette more than 30 minutes after awaking.
  4 mg lozenge for participants who usually smoke their first cigarette less than 30 minutes after awaking.
  Replace each forgone cigarette while abstinent with one lozenge. Use additional lozenges to combat cravings to smoke.
  Other Names: Commit Nicotine Lozenges

SUMMARY:
This study tests whether stopping smoking by gradually cutting down first is more or less successful than stopping abruptly. We hypothesize that stopping by gradually cutting down first will produce more abstinence than stopping abruptly.

DETAILED DESCRIPTION:
For cigarette smokers who intend to stop smoking, most treatment guidelines recommend abrupt cessation. There is evidence from some small studies that gradually reducing the number of cigarettes per day smoked may increase success in quitting. In this study, we will randomize smokers who want to quit smoking in the next 30 days to one of three groups: gradual reduction, abrupt cessation, and minimal intervention.

ELIGIBILITY:
Inclusion Criteria:

* Interested in quitting gradually
* At least 18 years old
* Daily cigarette smoker
* Smoke at least 15 cigarettes per day (CPD)
* No change greater than 20% in CPD in the last month
* Interested in quitting in next 30 days
* Must agree to not use non-cigarette tobacco during study
* No use of smoking cessation medication in last month
* Have phone with voice mail
* Willing to use nicotine lozenge
* No other person in household in study
* Fluent/literate in English

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Currently using medication for depression or asthma
* Heart disease requiring medication
* Heart attack in last month
* Irregular heartbeat
* High blood pressure not controlled by medication
* Stomach ulcers
* Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2006-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hughes, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont Human Behavioral Pharmacology Lab, Burlington, Vermont, United States

REFERENCES:
- [Result] Hughes JR, Solomon LJ, Livingston AE, Callas PW, Peters EN. A randomized, controlled trial of NRT-aided gradual vs. abrupt cessation in smokers actively trying to quit. Drug Alcohol Depend. 2010 Sep 1;111(1-2):105-13. doi: 10.1016/j.drugalcdep.2010.04.007. Epub 2010 May 26. PMID 20537810

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited using advertisements targeting smokers who wanted to quit smoking gradually. Advertisements were placed in newspapers in two cities in South Carolina and one city in New Mexico.
Pre-assignment Details: Enrolled sample size of 750; 4 were excluded because found to be ineligible after enrollment.
Groups:
- Gradual Reduction: Counseling of smokers to undergo gradual reduction in cigarettes per day prior to quit date
- Abrupt Cessation: Counseling of smokers to set a quit date and not change cigarettes per day prior to quit date
- Minimal Intervention: Minimal intervention to mimic intervention at a primary care office
Period: Set Quit Date
Arm/Group | Gradual Reduction | Abrupt Cessation | Minimal Intervention
Started | 297 | 299 | 150
Completed | 290 | 286 | 145
Not Completed | 7 | 13 | 5
Not completed — Lost to Follow-up | 7 | 13 | 5
Period: 6 Month Follow-up
Arm/Group | Gradual Reduction | Abrupt Cessation | Minimal Intervention
Started | 290 | 286 | 145
Completed | 227 | 237 | 118
Not Completed | 63 | 49 | 27
Not completed — Lost to Follow-up | 63 | 49 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gradual Reduction | Abrupt Cessation | Minimal Intervention | Total
Number analyzed (Participants) | 297 | 299 | 150 | 746
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 273 | 276 | 139 | 688
  >=65 years | 24 | 23 | 11 | 58
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (13) | 48 (12) | 47 (13) | 48 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 165 | 80 | 404
  Male | 138 | 134 | 70 | 342
Region of Enrollment [Number; unit: participants]
  United States | 297 | 299 | 150 | 746

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Prolonged Abstinence Through 6 Months Verified by Carbon Monoxide Measurement
Description: Number of participants with self-reported prolonged abstinence from cigarette smoking through 6 months of follow-up, verified by a breath carbon monoxide reading of less than 10 parts per million
Time Frame: 6 months
Population: This was an intent-to-treat analysis. Those who were lost to follow-up were assumed to not be abstinent from smoking at the time of the 6 month follow-up.
Measure: Number; unit: participants
Groups:
- Gradual Reduction: Counseling of smokers to undergo gradual reduction in cigarettes per day prior to quit date; nicotine lozenges were provided to aid reduction prior to the quit date and for use on and following the quit date.
- Abrupt Cessation: Counseling of smokers to set a quit date and not change cigarettes per day prior to quit date; nicotine lozenges were provided for use starting on the quit date.
- Minimal Intervention: Minimal intervention to mimic intervention at a primary care office; nicotine lozenges were provided for use starting on the quit date.
Arm/Group | Gradual Reduction | Abrupt Cessation | Minimal Intervention
Number analyzed (Participants) | 297 | 299 | 150
participants | 12 | 20 | 7
Statistical Analysis 1: Comparison: Gradual Reduction vs Abrupt Cessation vs Minimal Intervention; Null hypothesis: prolonged abstinence from smoking is the same for the three groups at 6 month follow-up Sample size was based on an assumption of 6 month abstinence of 25% in the gradual group, 15% in the abrupt group, and 10% in the minimal group. Sample sizes of 300, 300, and 150 for gradual, abrupt, and minimal provides 97% to detect a difference between the groups, with 2-sided alpha = 0.05; Test type: Superiority or Other; p = 0.30, Chi-squared — Statistical significance was determined by a two-sided p value less than 0.05; Degrees of freedom = 2
Statistical Analysis 2: Comparison: Gradual Reduction vs Abrupt Cessation; Test type: Superiority or Other; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.28 to 1.22] — The reported odds ratio represents the odds of 6 month prolonged abstinence in the gradual reduction group divided by the odds of 6 month prolonged abstinence in the abrupt cessation group

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Gradual Reduction | Abrupt Cessation | Minimal Intervention
Serious Adverse Events (participants affected / at risk) | 0/297 | 0/299 | 0/150
Other Adverse Events (participants affected / at risk) | 0/297 | 0/299 | 0/150

LIMITATIONS AND CAVEATS:
Our projected incidence of abstinence was higher than what was actually observed, leading to lower statistical power than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No